CLINICAL TRIAL: NCT02151487
Title: A Comparison of Ropivacaine Alone Versus Ropivacaine With Dexamethasone or Clonidine Versus a Combination of Ropivacaine, Dexamethasone, and Clonidine for Supraclavicular Brachial Plexus Block Using Ultrasound:A Prospective, Observer-blinded, Randomized Study
Brief Title: A Comparison of Ropivacaine Alone Versus Combination of Dexamethasone and Clonidine for Block
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Dawood Nasir, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: 102013-068
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Upper Extremity Surgery
Keywords: Supraclavicular block; Ropivacaine; Dexamethasone; Clonidine; Postoperative analgesia
MeSH Terms: interventions — Ropivacaine; Dexamethasone; Adjuvants, Pharmaceutic; Clonidine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Ropivacaine: Ropivacaine 0.5% 25 ml alone for supraclavicular block
  Interventions: Drug: Ropivacaine
- Ropivacaine and dexamethasone: 25 ml 0.5% ropivacaine + 4 mg dexamethasone
  Interventions: Drug: Ropivacaine and dexamethasone
- Ropivacaine and clonidine: 25 ml 0.5% ropivacaine + 100 mcg clonidine
  Interventions: Drug: Ropivacaine and clonidine
- Ropivacaine, dexamethasone and clonidine: 25 ml 0.5% ropivacaine + 4 mg dexamethasone + 100 mcg clonidine
  Interventions: Drug: Ropivacaine, dexamethasone and clonidine

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine alone
  Other Names: Noropin
  Groups: Ropivacaine
Drug: Ropivacaine and dexamethasone — Ropivacaine combination with dexamethasone
  Other Names: Noropin and adjuvant
  Groups: Ropivacaine and dexamethasone
Drug: Ropivacaine and clonidine — Ropivacaine combination with clonidine
  Other Names: Noropin and adjuvants
  Groups: Ropivacaine and clonidine
Drug: Ropivacaine, dexamethasone and clonidine — Ropivacaine combination with dexamethasone and clonidine
  Other Names: Noropin and adjuvants
  Groups: Ropivacaine, dexamethasone and clonidine

SUMMARY:
The aim of this randomized, observer-blinded study is to evaluate the postoperative analgesic efficacy of adding dexamethasone and clonidine to ropivacaine in supraclavicular nerve block. The investigators hypothesized that addition of dexamethasone and clonidine to ropivacaine would prolong the duration of analgesia in supraclavicular nerve block compared with ropivacaine alone.

DETAILED DESCRIPTION:
Subjects undergoing orthopedic surgery of upper extremities were randomized to be one of the three groups to receive supraclavicular nerve block with group 1: ropivacaine alone; group 2: ropivacaine and dexamethasone; group 3: ropivacaine and clonidine or group 4: ropivacaine and dexamethasone and clonidine combination.

Subjects were identified at the day surgery unit at Parkland hospital before the procedure and approached by their physician, the primary investigator, or research personnel for the consent for the study. If the subjects chooses and consents fully to participate, he or she was randomly assigned to receive one of the previously described local anesthetics for supraclavicular nerve block.

The following clinical outcomes were assessed for up to 24 hr: Duration of the block, onset of the block, postoperative pain scores, nausea, vomiting, and complications of peripheral nerve block. Pain was evaluated by using a linear 10-cm visual analog scale (VAS; 0=no pain, 10= worst imaginable pain) immediately before the block, 5, 10, 15 minutes and postoperatively on the arrival of Post Anesthesia Care Unit (PACU) within 15 minutes, discharge from the Day surgery Unit, and 24 hr. later at home via phone call visit.

Sensory and motor block in the related nerve dermatomes were assessed. Patient was instructed to document at what time did hand motion (finger movement) return and what time normal sensation return. Specific time for both events was sked to patient at phone call visit 24 hr later. Overall patient satisfaction was evaluated at the discharge from the day surgery and 24 hr after the block via phone visit.

At any point in which the patient is not experiencing pain relief after having received the injection, they were removed from the study and other anesthetic techniques will be applied to resolve their pain along with pharmacological management of their pain. Rescue antiemetic, which is standard of care, will be given to any patient who complains of nausea or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-80 years old
* Undergoing upper extremity surgery
* Receiving Supraclavicular block
* Receiving ropivacaine, ropivacaine adjuvants (dexamethasone, clonidine) for the supraclavicular nerve block.
* Able to give Informed consent

Exclusion Criteria:

* Age less than 18 and greater than 80 years
* Inability to understand the study procedures
* Significant respiratory dysfunction
* Preexisting neurologic deficits
* Allergy to local anesthetics
* A bleeding diathesis or on anticoagulants
* Systemic glucocorticoid use
* Refuse to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who scheduled to undergo upper extremity surgery requiring USSB for postoperative analgesia with ropivacaine alone or ropivacaine and adjuvants.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawood Nasir, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study takes place in routine clinical context. Subjects who received supraclavicular nerve block with ropivacaine alone or ropivacaine with adjuvants enrolled to the study.
Period: Overall Study
Arm/Group | Ropivacaine | Ropivacaine and Dexamethasone | Ropivacaine and Clonidine | Ropivacaine, Dexamethasone and Clonidine
Started | 27 | 27 | 20 | 23
Completed | 25 | 22 | 16 | 20
Not Completed | 2 | 5 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ropivacaine | Ropivacaine and Dexamethasone | Ropivacaine and Clonidine | Ropivacaine, Dexamethasone and Clonidine | Total
Number analyzed (Participants) | 27 | 27 | 20 | 23 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Participants were ambulatory cases and followed with 24 h phone call visit. Due to follow-up lost, analysis population is lower than overall population.
  years
    number analyzed (Participants) | 25 | 22 | 16 | 20 | 83
    (all) | 49 (16) | 43 (14) | 48 (11) | 50 (11) | 48 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Subjects were ambulatory surgery cases and followed via phone call visit 24 hours after discharge.
  Participants
    number analyzed (Participants) | 25 | 22 | 16 | 20 | 83
    Female | 10 | 13 | 8 | 10 | 41
    Male | 15 | 9 | 8 | 10 | 42

OUTCOME MEASURES:

1. Primary Outcome: Duration of the Sensorial Supraclavicular Block
Description: Duration of sensorial block defined as the time interval between subject admitted to the Post-Anesthesia Care Unit and the time the first pain medication taken at home
Time Frame: within 24-hr after surgery
Population: Participants received supraclavicular nerve block with ropivacaine alone and ropivacaine with adjuvants.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Ropivacaine | Ropivacaine and Dexamethasone | Ropivacaine and Clonidine | Ropivacaine, Dexamethasone and Clonidine
Number analyzed (Participants) | 25 | 22 | 16 | 20
hour | 13.4 (6) | 14 (6.6) | 17.4 (6) | 18.8 (6.2)

2. Secondary Outcome: Postoperative Analgesia
Description: Post-operative Visual Analog Pain (VAS) scores on the scale of 10 (0=no pain and 10=worse imaginary pain).
Time Frame: within 15 minutes at postanesthesia care unit (PACU) arrival
Population: Patients received supraclavicular nerve block with ropivacaine alone or ropivacaine with adjuvants. Postoperative pain was evaluated by using Visual Analog Pain Scores on the scale of 10 (0=no pain and 10-worse pain).
Measure: Median (Inter-Quartile Range); unit: score on a scale of 10
Arm/Group | Ropivacaine | Ropivacaine and Dexamethasone | Ropivacaine and Clonidine | Ropivacaine, Dexamethasone and Clonidine
Number analyzed (Participants) | 25 | 22 | 16 | 20
score on a scale of 10 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Following nerve block to postoperative 24 hour period.
Arm/Group | Ropivacaine | Ropivacaine and Dexamethasone | Ropivacaine and Clonidine | Ropivacaine, Dexamethasone and Clonidine
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 0/27 | 1/27 | 0/20 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ropivacaine (N=27) | Ropivacaine and Dexamethasone (N=27) | Ropivacaine and Clonidine (N=20) | Ropivacaine, Dexamethasone and Clonidine (N=23)
Shortness of breath (SOB) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Shortness of breath immediately after nerve block

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No